CLINICAL TRIAL: NCT03254953
Title: GoalTracker: Comparing Self-Monitoring Strategies for Weight Loss: Does Developing Mastery Before Tracking Diet Enhance Engagement?
Brief Title: GoalTracker: Comparing Self-Monitoring Strategies for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0822
Record Dates: First submitted 2017-08-07; First posted 2017-08-21 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Overweight; Weight Loss
Keywords: digital health; eHealth; technology; smartphone; obesity; overweight; weight loss; behavioral intervention; self-monitoring; tracking; engagement; adherence; weight change; e-mail; mobile application; goal setting; action plan; feedback; electronic health
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: 12-week randomized controlled trial to compare 3 self-monitoring approaches for weight loss in a digital health intervention for adults who are overweight or obese
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequential Intervention (Experimental): * in this Sequential eHealth intervention, participants are asked to self-monitor only their body weight for the first month, then for months 2 and 3 they will be asked to also self-monitor their diet
  * participants are asked to use the MyFitnessPal app for self-monitoring
  * given goal to lose 5% weight by end of intervention (3 months)
  * weekly personalized feedback via email
  * weekly skills training materials (behavioral modification lessons; tips on using different features of the app) via email
  * weekly action plans via email
  Interventions: Behavioral: self-monitoring of body weight; Behavioral: self-monitoring of diet; Behavioral: weekly personalized feedback + lessons + action plans
- Simultaneous Intervention (Experimental): * in this Simultaneous eHealth intervention, participants are asked to self-monitor both their body weight and diet for 3 months
  * participants are asked to use the MyFitnessPal app for self-monitoring
  * given goal to lose 5% weight by end of intervention (3 months)
  * weekly personalized feedback via email
  * weekly skills training materials (behavioral modification lessons; tips on using different features of the app) via email
  * weekly action plans via email
  Interventions: Behavioral: self-monitoring of body weight; Behavioral: self-monitoring of diet; Behavioral: weekly personalized feedback + lessons + action plans
- Control (diet-tracking only) (Experimental): * participants are asked to self-monitor their diet for 3 months
  * participants are asked to use the MyFitnessPal app for self-monitoring
  * given goal to lose 5% weight by end of intervention (3 months)
  Interventions: Behavioral: self-monitoring of diet

INTERVENTIONS:
Behavioral: self-monitoring of body weight — - weigh daily for 3 months and track their weight using the MyFitnessPal mobile app
  Arms: Sequential Intervention; Simultaneous Intervention
Behavioral: self-monitoring of diet — * track their diet (food and drinks) daily using the MyFitnessPal mobile app
  * when they are asked to track diet will vary based on the arm
Behavioral: weekly personalized feedback + lessons + action plans — - these are additional evidence-based intervention components
  Arms: Sequential Intervention; Simultaneous Intervention

SUMMARY:
This study is a randomized controlled trial that compares 3 self-monitoring approaches for weight loss. GoalTracker is a standalone, technology-based intervention using a commercial smartphone app (MyFitnessPal) and email.

The investigators hypothesize that the group that delays diet tracking and receives additional intervention components (weekly personalized feedback, skills training, and action plans) will have greater weight loss at the end of the 12-week intervention and at 6-month followup, compared to (a) an intervention group that simultaneously tracks weight and diet for all 12 weeks and receives the same additional components, and (b) a control group that tracks only diet.

DETAILED DESCRIPTION:
This study will examine whether a digital health intervention (GoalTracker) can promote weight loss among adults who are overweight or obese. Engagement in self-monitoring often declines over time, which is then associated with suboptimal weight loss. Finding ways to improve self-monitoring engagement, particularly in the first month of treatment, is needed. Promoting mastery, self-efficacy, and self-regulatory skills may help with maintaining high engagement.

The investigators aim to enroll 105 participants. All groups are asked to self-monitor daily on their smartphone using the free commercial mobile application MyFitnessPal over the course of the 12-week intervention.

Specifically, the study aims to...

1. Determine the effect of a Sequential self-monitoring intervention, compared to a Simultaneous self-monitoring intervention on weight change, caloric intake change, and proportion of individuals achieving 5% weight loss.
2. Determine the effect of the Sequential self-monitoring intervention, compared to the Control, on the same variables.
3. Compare self-monitoring engagement by intervention arm.
4. Examine the relation between self-monitoring engagement and weight loss.
5. Investigate theoretical mediators (self-efficacy, mastery, and self-regulation) on the relation between treatment arm and weight change.

ELIGIBILITY:
Inclusion Criteria:

* ages 21-65 years old
* Body Mass Index (BMI) 25-45 kg/m2
* interested in losing weight through dietary change
* current use of iPhone or Android smartphone
* current use of email address
* has daily access to a bathroom scale
* no recent weight loss (≥10 lbs) in the past 6 months
* able to read and write in English
* able to attend 3 in-person evaluation visits at Duke University in Durham, North Carolina over a 3-month period

Exclusion Criteria:

* current participation in another weight loss treatment
* currently pregnant or planning to become pregnant within study period, or < 1 year post-partum
* history of cardiovascular event, eating disorder, diabetes mellitus, hypothyroidism, cancer, end stage renal disease
* current uncontrolled hypertension
* use of the MyFitnessPal app to track food in the past 6 months
* Former or planned bariatric surgery
* current use of medication (e.g., lithium, steroids, anti-psychotics)
* use of weight loss medication in past 6 months
* profound cognitive, developmental, or psychiatric disorders or recent hospitalization in a psychiatric facility

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 1 month, 3 months
  Weight will be collected in kilograms using a calibrated digital scale

SECONDARY OUTCOMES:
Proportion of Individuals Achieving ≥ 5% Weight Loss | Baseline to 3 months
  Weight will be collected in kilograms using a calibrated digital scale
Change in Caloric Intake | Baseline, 3 months
  Caloric intake will will be assessed using the Automated Self-Administered 24-hour Dietary Intake Assessment (ASA24), an online dietary recall tool developed by the National Cancer Institute
Change in Weight at 6 Months | 6 months
  At 6-months (i.e., 3 months post-intervention), self-reported weight will be collected
Self-Monitoring Engagement | Baseline to 1-month and 3 months
  Frequency of self-monitoring weight and diet; Consistency of self-monitoring weight and diet
Self-Efficacy | Baseline, 1 month, 3 months
  Weight Efficacy Lifestyle Questionnaire (WEL) (20 items) will assess self-efficacy for eating. Separate surveys that were adapted will assess self-efficacy for self-monitoring of diet and weight.
Mastery | Baseline, 1 month, 3 months
  The Automaticity subscale of The Self-Report Habit Index (SRHI) will assess mastery of self-monitoring diet and weight (4 items each).
Self-Regulation | Baseline, 1 month, 3 months
  The Three Factor Eating Questionnaire-R18 (TFEQ-R18) (18 items) will assess self-regulation for controlled eating. Separate surveys that were adapted will assess self-regulation for self-monitoring of diet and weight.

OTHER OUTCOMES:
Physical Activity | Baseline, 3 months
  Paffenbarger Activity Questionnaire (7 items) will assess physical activity.
Sleep Quality | Baseline, 1 month, 3 months
  Medical Outcomes Study (MOS) Sleep (12 items) will assess sleep quality.
Perceived Stress | Baseline, 3 months
  Perceived Stress Scale (10 items)
Depressive Symptoms | Baseline, 1 month, 3 months
  Patient Health Questionnaire (PHQ-8) will assess depressive symptoms.
Health-Related Quality of Life | Baseline, 1 month, 3 months
  EuroQol-5 Dimension (EQ-5D) (5 items) will assess health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michele G Lanpher, MA, Principal Investigator — Duke University; Gary G Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
This data set is initially being used for the principal investigator's (Michele Lanpher) doctoral dissertation.

REFERENCES:
- [Derived] Patel ML, Hopkins CM, Brooks TL, Bennett GG. Comparing Self-Monitoring Strategies for Weight Loss in a Smartphone App: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Feb 28;7(2):e12209. doi: 10.2196/12209. PMID 30816851